CLINICAL TRIAL: NCT05837871
Title: Assessment of Genetic and Haematological Modifiers of Disease Severity Among Patients With Sickle Cell Disease (SCD) in Kaduna State, Northern Nigeria
Brief Title: Genetic and Haematological Modifiers of SCD Severity in Kaduna State, Northern Nigeria
Acronym: SCA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmadu Bello University Teaching Hospital (Other)
Collaborators: Cyprus Institute of Neurology and Genetics (Other)
Responsible Party: Principal Investigator, Bello Jamoh Yusuf, Dr, Ahmadu Bello University Teaching Hospital
Other Study IDs: ABUTH
Record Dates: First submitted 2023-03-14; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Sickle Cell Disease
Keywords: Genetics; Haematological parameters; Modifiers; Sickle Cell Disease; Kaduna, Nigeria; Assessment
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole peripheral blood sample and Extracted DNA from peripheral mononuclear cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross sectional arm: Patients with Sickle Cell Anaemia aged 2 to 18 years. Assessed for clinical severity, Complete Blood Count, foetal haemoglobin and Haemoglobin Haplotype
- Longitudinal arm: * Patients with Sickle Cell Anaemia recruited at 9 months of age then followed up at 12 months, 18 months and 24 months.
  * Assessed for clinical severity, Complete Blood Count, foetal haemoglobin and Haemoglobin Haplotype
  * Both parents assesed for Haemoglobin Haplotype
  * Genotype - Haplotype assessment to be carried out

SUMMARY:
This study is aimed to assess the genetic and haematological modifiers of disease severity among patients with Sickle Cell Disease (SCD) in Kaduna State, northern Nigeria. It is composed by two separate study designs: a cross-sectional study and a longitudinal study.

The cross-sectional study will evaluate clinical and laboratory parameters in paediatric Sickle Cell Anaemia (SCA) patients (ages 2-18 years) in steady state and during Vaso-Occlusive Crisis (VOCs) to determine the parameters that can be used as a guide to monitor the course of the disease towards early recognition and management of sickle cell crises. In addition, the study will explore genotype-phenotype correlations in SCA patients by targeted Next-Generation Sequencing (NGS) of genetic modifiers for haemoglobinopathies.

The longitudinal study will collect clinical and laboratory data over time for a paediatric cohort of SCD patients (9 months old; followed up to 2 years of age) and parental samples will be collected to determine the βS-globin haplotype in family trios. The aim is to determine the temporal relationships among foetal haemoglobin (HbF) levels, haematological parameters and frequency of sickle cell crises in SCD patients in relation to the type of the βS-globin haplotype and the sickle genotype. In addition, samples collected at 24 months of age will also be analysed by NGS to identify genetic modifiers of clinical manifestations and severity of SCA.

Participants from the following centre will be involved: Ahmadu Bello University Teaching Hospital (ABUTH) Zaria. Consent from all the study parents/legally designated representatives as well as assent from minors will be sought. Consent for genetic analyses will be sought as well. Clinical and haematological analyses will be performed at ABUTH while genetic analyses will be performed at the Cyprus Institute of Neurology and Genetics (CING).

DETAILED DESCRIPTION:
Sickle cell anaemia (SCA) is a multisystem disorder with massive medical, social and financial implications worldwide. It is caused by a single mutation in the β-globin gene (β6 Glu>Val), which leads to the production of abnormal sickle haemoglobin (HbS). Africa is the major origin of the sickle (βS) mutation, which occurs on diverse genetic haplotype backgrounds. SCA has a Mendelian pattern of inheritance (βS gene homozygosity, i.e. HbSS). Although all SCA patients share the same genetic mutation, the disease exhibits wide heterogeneity in clinical expression, which can be explained by both environmental and genetic factors. The environmental factors include infections, trauma, climate (temperature and humidity) and air quality, as well as socioeconomic factors, many of which are controllable. The genetic factors, on the other hand, cannot be controlled. The best-characterized genetic factors include variants in the genes associated with foetal haemoglobin (HbF) production, co-inheritance of alpha-thalassaemia, sickle genotype, and the type of βS-globin haplotype. The role of other potential genetic modifiers is less clear, particularly with regards to sickle cell disease related organ damage (e.g., risk for stroke, haemolysis, and acute chest syndrome.

Understanding the molecular basis of clinical heterogeneity and disease severity for SCA can have direct clinical applications for prognosis via risk stratification of patients, also facilitating the use of personalized, targeted therapeutic interventions. As a turning-point in genomics, the advent of high-throughput sequencing and whole-genome analysis has made it feasible to discover hitherto unsuspected variants that could add to current understanding of genotype-phenotype relationships in SCA. The identification of modifying genetic variants might suggest new prognostic and/or therapeutic targets for investigation towards improved patient management and treatment.

ELIGIBILITY:
Inclusion Criteria:

* (i) Paediatric patients (ages 2-18 years) with known HbSS genotype from case records. They will be recruited during routine visits at the haematology clinics.

(ii) Patients in steady-state and in sickle cell crisis.

* Patients will be considered to be in steady-state if they are in a period free of crisis extending from at least three weeks since the last clinical event and three months or more since the last blood transfusion, to at least one week before the start of a new clinical event.
* Patients will be considered to be in sickle cell crisis (i.e. vaso-occlusive crisis, VOC) if they are known to have SCD, together with bone or joint pain, or multiple sites of pain, necessitating hospital admission and analgesic administration.

(iii) Paediatric patients enrolled at 3 months of age with SCD diagnosed during newborn screening and followed over time at 6 months, 9 months, 12 months and 24 months of age.

(iv) A written informed consent signed by all participants and/or parents/legally designated representatives is required to be recruited.

Exclusion Criteria:

* (i) Subjects with overt features of significant co-morbidities like malignancies, malnutrition, congenital deficiencies or severe infections.

Ages: 9 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Sickle Cell Anaemia attending Clinics in Ahmadu Bello University Teaching Hospital, Zaria Nigeria.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Cross sectional arm | 3 months
  Subjects with Sickle Cell disease (n=200), aged 2 - 18 years will be recruited for this arm of the study
  * Clinical severity using the severity index developed by van den Tweel et al in PMID 20806231
  * Complete blood count using Coulter Haematology Auto-analyzer: WBC (10^9/L), RBC (10^12/L), Hb (g/L), HCT (%), PLT (10^9/L), MCV (fl), MCH (pg), MCHC (g/L)
  * Foetal haemoglobin using HPLC - 10 machine: (%)
  * Hemoglobin haplotype using a SNPs test [RFLP-PCR] to determine beta S-globin haplotypes

SECONDARY OUTCOMES:
Longitudinal arm | 18 months
  Subjects with SCD (n=200) at 9 months of age will be recruited and followed up at 12months, 18months and 24months
  * Clinical severity index developed by van den Tweel et al in PMID 20806231, will be assessed at each follow-up contact.
  * Complete blood count using Coulter Haematology Auto-analyzer: WBC (10^9/L), RBC (10^12/L), Hb (g/L), HCT (%), PLT (10^9/L)
  * Foetal haemoglobin using HPLC - 10 machine: (%)
  * Hemoglobin analysis using a SNPs test [RFLP-PCR] to determine beta S-globin haplotype.
  * Spatial relationship of parameters (Blood counts, Severity scores, Level of HbF) will be correlated (using Spearman or Pearson), depending on normality of distribution of the data.
  * Parental samples (of each subject above) will be obtained for genomic characterization of Beta S globin gene in family trios.
  * Chi-squrared test or Wilcoxon's (as appropriate) will be used to associate certain outcome measures (e.g., HbF, severity) with specific beta S globin gene haplotypes

IPD SHARING:
Plan to Share IPD: Yes
IPD will be freely shared with researchers and students
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available in 2 years with limitless access